CLINICAL TRIAL: NCT00713687
Title: Sequential Combination of Chemotherapy With Gemcitabine/Oxaliplatin and Photodynamic Therapy in Advanced Cholangiocarcinoma
Brief Title: Gemcitabine/Oxaliplatin and Photodynamic Therapy in Cholangiocarcinoma
Acronym: GemOx-PDT
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: recruiting failed
Sponsor: Technical University of Munich (Other)
Collaborators: Münchner Studienzentrum (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEM-658-EBE-0024-I; EudraCT-Nr.: 2008-001560-37
Record Dates: First submitted 2008-07-07; First posted 2008-07-11 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2008-07

CONDITIONS: Cholangiocarcinoma
Keywords: photodynamic therapy; PDT; gemcitabine; oxaliplatin; cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Gemcitabine; Oxaliplatin; Photochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Treatment by combination of photodynamic therapy and chemotherapy
  Interventions: Drug: Gemcitabine, Oxaliplatin, Photodynamic therapy (Photosan®)

INTERVENTIONS:
Drug: Gemcitabine, Oxaliplatin, Photodynamic therapy (Photosan®) — 1. Photodynamic therapy (PDT) after successful drainage:
     Photosan® 2 mg/kg i.v. 48 hrs before laser activation
  2. 9 cycles of GemOx chemotherapy (start 4 weeks after PDT):
     * Gemcitabine 1000 mg/m² 100 min infusion on day 1 of chemotherapy
     * Oxaliplatin 100 mg/m² 2h infusion on day 2 of chemotherapy
     * iteration every 14 days
     * afterwards 4 weeks intermission
  3. Iteration of 1. and 2. in case of good compatibility
  Other Names: No other names

SUMMARY:
In patients with cholangiocarcinoma therapeutic effects have been reported for Gemcitabine/Oxaliplatin. Furthermore, photodynamic therapy (PDT) has significantly improved patients survival in two randomised trials. PDT induces tumor necrosis only in an area of few millimetres, while tumor parts which are located beyond this area remain untreated. An additive effect could result from PDT as a local therapy in combination with systemic chemotherapy.

DETAILED DESCRIPTION:
Patients entered in the study receive a sequential therapy consisted of photodynamic therapy followed by systemic chemotherapy (Gemcitabine/Oxaliplatin) 4 weeks later. Systemic chemotherapy every 2 weeks is scheduled 9 times in each cycle. Thereafter, another cycle of PDT followed by chemotherapy is intended.

ELIGIBILITY:
Inclusion Criteria:

* Histologic/cytologic verified cholangiocarcinoma or cholangiocarcinoma-typical findings in >= 2 diagnostic methods
* Bile duct stenoses which are technically successful treated with biliary drainage
* Irresectability/inoperability
* Karnofsky-Index >= 60%
* Age >= 18
* Written consent

Before chemotherapy:

* Bilirubin <= 5 mg/dl
* GOT/GPT < 5x upper standard
* Creatinine < 2x upper standard
* Thrombocytes > 100 G/l
* Neutrophils > 2,00 G/l
* Haemoglobin > 9 g/dl
* No occurence of complications during endoscopic procedures (abscess, bilioma, cholecystitis, cholangitis, pancreatitis, biliary leakage)

Exclusion Criteria:

* Implantation of a metal stent in the bile duct
* Previous PDT or chemotherapy
* Neoplasia
* Porphyria
* Pregnant or breastfeeding women
* Women of childbearing age and potent men who are not using highly effective contraceptives

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-08; Study Completion 2011-12

PRIMARY OUTCOMES:
Progression free survival 6 months after study start | 6 months after study start

SECONDARY OUTCOMES:
Progression free survival 12 months after study start Progression free interval Overall survival Life quality | Until 12 months after study start

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Ebert, Prof. Dr., Principal Investigator — Head of the gastroenterological department of the Klinikum rechts der Isar; Roland M. Schmid, Prof. Dr., Study Chair — Head of the gastroenterological department of the Klinikum rechts der Isar
Locations (1):
- Technical University of Munich at the Klinikum rechts der Isar II. Medizinische Klinik Ismaninger Str. 22, Munich, Germany

REFERENCES:
- [Background] Rajagopalan V, Daines WP, Grossbard ML, Kozuch P. Gallbladder and biliary tract carcinoma: A comprehensive update, Part 1. Oncology 2004;18:889-896. Patel T. Cholangiocarcinoma. Nat Clin Pract Gastroenterol Hepatol 2006;3:33-42. de Groen PC, Gores GJ, LaRusso NF, Gunderson LL, Nagorney DM. Biliary tract cancers. N Engl J Med. 1999;341:1368-1378. Eckel F, Schmid RM. Chemotherapy in advanced biliary tract carcinoma: a pooled analysis of clinical trials. Br J Cancer 2007;96:896-902. Ortner ME, Caca K, Berr F, Liebetruth J, Mansmann U, Huster D, Voderholzer W, Schachschal G, Mössner J, Lochs H. Successful photodynamic therapy for nonresectable cholangiocarcinoma: a randomized prospective study. Gastroenterology 2003;125:1355-1363. Zoepf T, Jakobs R, Arnold JC, Apel D, Riemann JF. Palliation of nonresectable bile duct cancer: improved survival after photodynamic therapy. Am J Gastroenterol 2005;100:2426-2430. Wiedmann M, Caca K, Berr F, Schiefke I, Tannapfel A, Wittekind C, Mössner J, Hauss J, Witzigmann H. Neoadjuvant photodynamic therapy as a new approach to treating hilar cholangiocarcinoma: a phase II pilot study. Cancer. 2003;97:2783-2790. Dougherty TJ, Gomer CJ, Henderson BW, Jori G, Kessel D, Korbelik M, Moan J, Peng Q. Photodynamic therapy. J Natl Cancer Inst. 1998;90:889-905. Gollnick SO, Vaughan L, Henderson BW. Generation of effective antitumor vaccines using photodynamic therapy. Cancer Res 2002;62:1604-1608. Wiedmann M, Berr F, Schiefke I, Witzigmann H, Kohlhaw K, Mössner J, Caca K. Photodynamic therapy in patients with non-resectable hilar cholangiocarcinoma: 5-year follow-up of a prospective phase II study. Gastrointest Endosc 2004;60:68-75.